CLINICAL TRIAL: NCT03788837
Title: " ILOPROST for Treatment of Septic Shock With Persistent Microperfusion Defects ", a Double-blind, Randomized Controlled Trial:The I-MICRO Trial
Brief Title: ILOPROST in Septic Shock With Persistent Microperfusion Defects (I-MICRO)
Acronym: I-MICRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P170924J
Record Dates: First submitted 2018-11-20; First posted 2018-12-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock Hyperdynamic
Keywords: Microcirculatory defects; hemodynamic macroparameters; mottling; Septic shock; SOFA score
MeSH Terms: conditions — Shock, Septic | interventions — Iloprost; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous ILOPROST (Experimental): a first dose of ILOPROST of 0.5ng/kg/ min with increments every 30 minutes up to a maximum of 1,5 ng/kg/min for 48h
  Interventions: Drug: ILOPROST
- Intravenous Placebo (Placebo Comparator): Treatment with intravenous NaCl 0.9% therapy with incremental infusion rate every 30 minutes for 48h
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: ILOPROST — The patient will receive treatment with intravenous ILOPROST therapy at a dose of 0.5ng/kg/min with increments of 0.5 ng/kg/min every 30 minutes up to a maximum posology of 1,5 ng/kg/min for 48h.
  Other Names: 50 microgrammes /0,5 ml vials
  Arms: intravenous ILOPROST
Drug: NaCl — The patient will receive treatment with intravenous NaCl 0.9% (placebo-double blinded) with increments of infusion rate every 30 minutes for 48h
  Other Names: (Saline 0.9%)
  Arms: Intravenous Placebo

SUMMARY:
Septic shock remains a major cause of death in critically ill patients. Alterations in microcirculation have long been proposed as a key pathophysiological factor of organ dysfunction and death in septic shock patients. Persistence of mottling, prolonged skin recoloration time and cyanosis of the extremities are the easily and frequently observed manifestations of these microcirculatory disorders. Ilomedin is a prostaglandin analog with a potent vasodilatory effect together with anti-thrombotic properties (inhibition of platelet aggregation) preferentially at the microcirculatory level. An increase in cardiac output with increased arterial oxygen delivery has been observed in clinical and preclinical studies with no episodes of hypotension. Improvement in mesenteric perfusion has moreover been observed in experimental sepsis using Ilomedin. Our group has furthermore reported that administration of Ilomedin in patients with refractory septic shock (peripheral hypoperfusion) resulted in a rapid and sustained improvement in peripheral perfusion. Altogether, Ilomedin may prevent or improve recovery of organ dysfunction in septic shock patients through recruitment of the microcirculation and, thereby, ultimately improve outcome.

DETAILED DESCRIPTION:
In the 32 participating centers: patients with septic shock and persistent peripheral hypoperfusion despite hemodynamic optimization (skin mottling and/or finger skin recoloration time > 3sec, and/or knee skin recoloration time > 4sec), after 6 to 24 hours of norepinephrine onset will be eligible for randomization.

Patients fulfilling the eligibility criteria will be included and randomized by the intensivist in two groups:

*Experimental group: The patient will receive treatment with intravenous Iloprost (blinded) therapy at a dose of 0.5 ng/kg/min with increments of 0.5 ng/kg/min every 30 minutes up to a maximum posology of 1.5ng/kg/min for 48h.

Placebo group: The patient will receive treatment with intravenous NaCl 0.9% (placebo-double blinded) therapy at a dose of 0.5ng/kg/min with increments of 0.5 ng/kg/min every 30 minutes according to body weight with a maximum posology of 1,5 ng/kg/min for 48h.

Primary outcome will be Delta Sequential Organ Failure Assessment (SOFA) score between infusion onset and day 7.

*within the 12 first hours after randomization : blood samples : 15 ml of blood will be collected at the same time as the sample routinely collected, within the 12 first hours after randomization in ICU, when the patients are perfused.

The blood will be drawn and worked as follows:

* 2 x EDTA tubes of 5 ml : After centrifugation each tube will be directly divided into 4 aliquots of 500 µL (8 aliquots per patient)
* 1 x aprotinine tube of 5 ml : After centrifugation, it will be directly divided into 4 aliquots of 500 µL

The aliquots previously will be stored locally, and will be transported to the "Centre de Ressources Biologiques" (CRB) of the Lariboisière Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Signed informed consent or inclusion under the emergency provisions of the law (Article L1122 -1-3 of the PHC / modified by Order n°2016-800 of June 16 2016 - art. 2).
* Patients with septic shock defined by the third international definition:

  * suspected or proven infection,
  * and organ dysfunction defined by an acute change in total SOFA score >or=2
  * and persistent hypotension requiring vasopressor treatment to maintain mean arterial pressure > 65 mmHg despite standard of care hemodynamic optimization
  * and serum lactate level > 2 mmol/L despite standard of care hemodynamic optimization
  * and persistence of peripheral hypoperfusion (skin mottling and/or finger skin recoloration time > 3sec, and/or knee skin recoloration time > 4sec) despite standard of care hemodynamic optimization
  * Within 6 to 24 hours after norepinephrine onset

Exclusion Criteria:

* Refusal to participate in the study
* Pregnancy, breastfeeding
* Hypersensitivity to Ilomedin or to any of the excipients.
* Conditions where the hemorrhagic risk may be increased due to the effects of Ilomedin on platelets (i.e., evolving hemorrhage, trauma, intracranial hemorrhage, active gastric ulcer).
* Platelet count < 10000 /mm3
* unstable angina.
* severe cardiac rhythm disorders since Norepinephrine onset
* severe hypoxemia (PaO2/FiO2 <100)
* myocardial infarction in the last 6 months
* lack of Social Insurance
* persons deprived of liberty
* persons of a protective measure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Delta (Sequential Organ Failure Assessment (SOFA)) score between infusion onset and day 7. SOFA score assesses organ failure (respiratory, hemodynamics, liver, coagulation, neurological and kidney) in ICU patients. | 7 days after randomisation
  SOFA and Delta SOFA calculation will be performed by the Intensivist. Patients deceased before day 7 will be attributed a maximum SOFA score.
  SOFA score range from 0 (no organ failure) to a maximum of 24 (worst SOFA score).

SECONDARY OUTCOMES:
Mean SOFA score during the first 7 days after randomization | 7 days after randomization
  SOFA and Delta SOFA calculation will be performed by the Intensivist.
Number of survival days outside ICU in the 28 days post randomization | Between ICU discharge and day 28
  It will be calculated by the number of days between ICU discharge and day 28 in survivors of ICU stay.
Number of ventilation-free survival days in the 28 days post randomization | Between randomization and day 28.
  It will be calculated as the number of survival days without mechanical ventilation
Number of renal replacement therapy-free survival days in the 28 days post randomization - | Between randomization and day 28.
  It will be calculated as the number of survival days without renal replacement therapy
Number of vasopressor-free survival days in the 28 days post randomization | Between randomization and day 28.
  It will be calculated as the number of survival days without vasopressor therapy
Molting score at day 1 after randomization. | At day 1 after randomization
  In order to identifying and quantifying microcirculatory dysfunction in septic shock. A picture of patient's knees will be taken.
  Molting score range from 0 to a maximum of 5 :
  0. - No mottling
  1. - Coin sized mottling area on the knee.
  2. - To the superior area of the knee cap.
  3. - Mottling up to the middle thigh
  4. - Mottling up to the fold of the groin
  5. - Severe mottling that extends beyond the the groin.
Conservation of plasma for future biological measurements | within 10 years after the end of the study.
  15 ml of blood will be collected at the same time as the sample routinely collected, within the 12 first hours after randomization, when the patients are perfused.
Microcirculation | At the baseline, and between day 2 and day 7
  Monitoring of microcirculation using non-invasive monitoring devices including: photoplethysmography,cutaneous Doppler coupled with iontophoresis, near-infrared spectroscopy, videomicroscopy, tissular PCO2, urethral photoplethysmography, perfusion index using phtoplethysmography
mortality | At day 28

CONTACTS AND LOCATIONS:
Overall Officials: François DEPRET, MD, Principal Investigator — APHP-Hôpital saint Louis; Matthieu LEGRAND, MD,PhD, Study Director — APHP-Hôpital saint Louis
Locations (1):
- Departement of Anesthesiology, Critical Care and Burn Unit; Saint-Louis hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Backer D, Donadello K. Assessment of microperfusion in sepsis. Minerva Anestesiol. 2015 May;81(5):533-40. Epub 2014 Jun 19. PMID 24941897
- [Background] Ait-Oufella H, Lemoinne S, Boelle PY, Galbois A, Baudel JL, Lemant J, Joffre J, Margetis D, Guidet B, Maury E, Offenstadt G. Mottling score predicts survival in septic shock. Intensive Care Med. 2011 May;37(5):801-7. doi: 10.1007/s00134-011-2163-y. Epub 2011 Mar 4. PMID 21373821
- [Background] Muller B, Schmidtke M. Microvascular effects of iloprost in the hamster cheek pouch. Adv Prostaglandin Thromboxane Leukot Res. 1987;17A:455-8. PMID 2444080
- [Background] Johannes T, Ince C, Klingel K, Unertl KE, Mik EG. Iloprost preserves renal oxygenation and restores kidney function in endotoxemia-related acute renal failure in the rat. Crit Care Med. 2009 Apr;37(4):1423-32. doi: 10.1097/CCM.0b013e31819b5f4e. PMID 19318827
- [Background] Hoeper MM, Gall H, Seyfarth HJ, Halank M, Ghofrani HA, Winkler J, Golpon H, Olsson KM, Nickel N, Opitz C, Ewert R. Long-term outcome with intravenous iloprost in pulmonary arterial hypertension. Eur Respir J. 2009 Jul;34(1):132-7. doi: 10.1183/09031936.00130408. Epub 2009 Feb 27. PMID 19251782
- [Background] Lara B, Enberg L, Ortega M, Leon P, Kripper C, Aguilera P, Kattan E, Castro R, Bakker J, Hernandez G. Capillary refill time during fluid resuscitation in patients with sepsis-related hyperlactatemia at the emergency department is related to mortality. PLoS One. 2017 Nov 27;12(11):e0188548. doi: 10.1371/journal.pone.0188548. eCollection 2017. PMID 29176794
- [Background] Depret F, Sitbon A, Soussi S, De Tymowski C, Blet A, Fratani A, Legrand M. Intravenous iloprost to recruit the microcirculation in septic shock patients? Intensive Care Med. 2018 Jan;44(1):121-122. doi: 10.1007/s00134-017-4935-5. Epub 2017 Sep 18. No abstract available. PMID 28921126
- [Derived] Legrand M, Jullien E, Kimmoun A, Geri G, Ait-Oufella H, Abrard S, Gaugain S, Bounes F, Guerci P, Pottecher J, Jamme M, Poncelin de Raucourt Y, Barraud D, Constantin JM, Juguet W, Lasocki S, Sonneville R, Audibert J, Plantefeve G, Ellrodt O, Fedou AL, Leone M, Lefebvre L, Auvet A, Chen D, Vicaut E, Depret F; I-MICRO Trial Investigators. Iloprost for the Treatment of Severe Septic Shock with Persistent Hypoperfusion: A Double-Blind, Randomized Controlled Trial. Am J Respir Crit Care Med. 2025 Jul;211(7):1211-1219. doi: 10.1164/rccm.202410-1924OC. PMID 40387381
- [Derived] Legrand M, Oufella HA, De Backer D, Duranteau J, Leone M, Levy B, Rossignol P, Vicaut E, Depret F; I-MICRO trial investigators. The I-MICRO trial, Ilomedin for treatment of septic shock with persistent microperfusion defects: a double-blind, randomized controlled trial-study protocol for a randomized controlled trial. Trials. 2020 Jul 1;21(1):601. doi: 10.1186/s13063-020-04549-y. PMID 32611377